CLINICAL TRIAL: NCT00942461
Title: Contribution to the Study of Inflammatory Response in Laparoscopic vs Open Colon Cancer Surgery
Brief Title: Inflammatory Response in Laparoscopic and Open Colectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: G. Hatzikosta General Hospital (Other)
Collaborators: University of Ioannina (Other)
Responsible Party: Konstantinos E. Tsimogiannis, MD, G. Hatzikosta General Hospital, Ioannina, Greece
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: GH-1948-04; GHDS-12345-4
Record Dates: First submitted 2009-07-20; First posted 2009-07-21 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Colorectal Cancer
Keywords: a-defensins; TLRs; Inflammatory Cytokines; CRP; No metastases; No other obvious inflammation; No chronic diseases
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Surgery group (Active Comparator): Group of patients that are operated with laparoscopic approach
  Interventions: Procedure: Laparoscopic colectomy
- Open surgery Group (Active Comparator): Group of patients operated with open approach
  Interventions: Procedure: Open colectomy

INTERVENTIONS:
Procedure: Laparoscopic colectomy — Laparoscopic colectomy. Epidural anaesthesia used
  Arms: Laparoscopic Surgery group
Procedure: Open colectomy — Open colectomy. Epidural anaesthesia used
  Arms: Open surgery Group

SUMMARY:
This study is designed to measure and compare the inflammatory response in laparoscopic and open colon cancer surgery

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer

Exclusion Criteria:

* metastases
* stage 4 colorectal cancer
* recurrent disease
* chronic diseases
* obvious inflammatory condition

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Inflammatory reaction of the patients organism in laparoscopic vs open colorectal surgery for cancer | preoperative, intraoperative, 6h postop, 24h postop

CONTACTS AND LOCATIONS:
Locations (1):
- G Hatzikosta General Hospital, Ioannina, Greece

REFERENCES:
- [Derived] Tsimogiannis KE, Tellis CC, Tselepis AD, Pappas-Gogos GK, Tsimoyiannis EC, Basdanis G. Toll-like receptors in the inflammatory response during open and laparoscopic colectomy for colorectal cancer. Surg Endosc. 2012 Feb;26(2):330-6. doi: 10.1007/s00464-011-1871-2. Epub 2011 Sep 5. PMID 21898023
- [Derived] Tsimogiannis KE, Telis K, Tselepis A, Pappas-Gogos GK, Tsimoyiannis EC, Basdanis G. Alpha-defensin expression of inflammatory response in open and laparoscopic colectomy for colorectal cancer. World J Surg. 2011 Aug;35(8):1911-7. doi: 10.1007/s00268-011-1140-5. PMID 21567262